CLINICAL TRIAL: NCT03186079
Title: Efficacy of Chinese Herbal Medicine Xiaojidaozhi Decoction in the Treatment of Childhood Functional Constipation: a Double Blind, Randomized and Placebo-controlled Trial
Brief Title: Efficacy of Chinese Herbal Medicine Xiaojidaozhi Decoction in the Treatment of Childhood Constipation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Shucheng Zhang, Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A333-2
Record Dates: First submitted 2017-06-04; First posted 2017-06-14 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Constipation; Chinese Herbal Medicine
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xiaojidaozhi Decoction (Active Comparator): Xiaojidaozhi Decoction and Fiberform and Toilet training are used for treatment of childhood Constipation
  Interventions: Drug: Xiaojidaozhi Decoction; Drug: Fiberform; Behavioral: Toilet training
- non-Xiaojidaozhi Decoction (Placebo Comparator): Placebo and Fiberform and Toilet training are used for treatment of childhood Constipation
  Interventions: Drug: Placebo; Drug: Fiberform; Behavioral: Toilet training

INTERVENTIONS:
Drug: Xiaojidaozhi Decoction — Mixture of twelve Chinese herbal medicines granule
  Other Names: XJD
  Arms: Xiaojidaozhi Decoction
Drug: Placebo — Mixture of 10% Chinese herbal medicines granule and 90% artificial gum
  Other Names: Placebos
  Arms: non-Xiaojidaozhi Decoction
Drug: Fiberform — Fiberform is a low-phytate wheat fibre which can increase the gastrointestinal motility.
Behavioral: Toilet training — Toilet training has been considered a routine method in treatment of constipation

SUMMARY:
Constipation is the most common complaint in childhood gastrointestinal disease,affecting an estimated 20% of the global children.The treatment strategies consist of diet control,behavioural intervention and oral and sometimes rectal laxatives. Given higher success rate and fewer side effects,the laxative PEG3350 has been considered the first choice in childhood constipation.However, effectiveness of PEG 3350 laxative is not lasting, additional treatment interventions are still necessary.With an unsatisfactory response to current treatments, many patients seek help from Chinese Herbal Medicine.In view of the traditional theory, childhood constipation is derived from weakness of gastric and splenic function.The functional weakness is characterized by food stagnation and further pathological heat accumulation in the gastrointestine. The food stagnation can slow the gastrointestinal motility while heat causes constipation by drying the intestines and their content. Therefore, the therapeutic principles and practices for childhood constipation must focus on the pathophysiological basis accordingly. In the documented traditional medicine dictionary(Pi Wei Lun), Xiaojidaozhi Decoction is well described in improving the gastric and splenic function, eliminating food stagnation and removing pathological heat accumulation, and it has always been used in treatment of constipation throughout Asia since the first description in Pi Wei Lun in 1249. It comprises twelve herbs. Through the combined action of these herbs, Xiaojidaozhi Decoction can increase fluid in the intestines and facilitate the gastrointestinal motility, relieving the symptoms of constipation. Despite of the long history of successful use of Xiaojidaozhi Decoction in childhood constipation, a large randomized placebo-controlled trial is still not available.The aim of this study was to explore the clinical efficacy and safety of Chinese herbal medicine Xiaojidaozhi Decoction in the treatment of childhood constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of childhood constipation
2. Criteria of constipation meets the Rome IV criteria(H3a)
3. Must be able to swallow capsules

Exclusion Criteria:

1. Digestive tract diseases
2. Neurologic diseases
3. Endocrine diseases
4. Metabolic diseases
5. Gastrointestinal surgery
6. Using drugs which can take impact on bowl motility

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Percentage of overall efficacy | week 8(end of treatment)
  Efficacy is ranked as cured, improved, same/worse
Percentage of overall efficacy | week 20(end of follow-up)
  Efficacy is ranked as cured, improved, same/worse
Baseline of constipation score in the beginning of treatment | beginning of treatment(baseline)
  Constipation is evaluated and scored on the related symptoms of stool frequency, appearance,consistency and incontinence
Change of constipation score from the baseline in the end of treatment | week 8(end of treatment)
  Constipation is evaluated and scored on the related symptoms of stool frequency, appearance,consistency and incontinence
Change of constipation score from the baseline in the end of follow-up | week 20(end of follow-up)
  Constipation is evaluated and scored on the related symptoms of stool frequency, appearance,consistency and incontinence

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Within week 20(end of follow-up)
  The adverse events reported in treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Voskuijl W, de Lorijn F, Verwijs W, Hogeman P, Heijmans J, Makel W, Taminiau J, Benninga M. PEG 3350 (Transipeg) versus lactulose in the treatment of childhood functional constipation: a double blind, randomised, controlled, multicentre trial. Gut. 2004 Nov;53(11):1590-4. doi: 10.1136/gut.2004.043620. PMID 15479678
- [Background] Tran LC, Di Palma JA. Lack of lasting effectiveness of PEG 3350 laxative treatment of constipation. J Clin Gastroenterol. 2005 Aug;39(7):600-2. doi: 10.1097/01.mcg.0000170769.67320.47. PMID 16000928
- [Background] Cheng CW, Bian ZX, Zhu LX, Wu JC, Sung JJ. Efficacy of a Chinese herbal proprietary medicine (Hemp Seed Pill) for functional constipation. Am J Gastroenterol. 2011 Jan;106(1):120-9. doi: 10.1038/ajg.2010.305. Epub 2010 Nov 2. PMID 21045817
- [Derived] Qiao L, Wang LJ, Wang Y, Chen Y, Zhang HL, Zhang SC. A Randomized, Double-Blind, and Placebo-Controlled Trial of Chinese Herbal Medicine in the Treatment of Childhood Constipation. Clin Transl Gastroenterol. 2021 May 3;12(5):e00345. doi: 10.14309/ctg.0000000000000345. PMID 33938874